CLINICAL TRIAL: NCT01538017
Title: Comparing Injectable Collagenase (CI) and Percutaneous Needle Fasciotomy (PNF) for Dupuytren's Contracture (DC) Affecting Proximal Interphalangeal Joints (PIP). A Randomised Controlled Trial
Brief Title: Injectable Collagenase and Percutaneous Needle Fasciotomy for Dupuytren's Contracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeppe Lange, MD (Other)
Responsible Party: Sponsor-Investigator, Jeppe Lange, MD, M:D:, Regionshospitalet Silkeborg
Organization: Regionshospitalet Silkeborg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-20110233
Record Dates: First submitted 2012-02-18; First posted 2012-02-23 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Dupuytrens Contracture
MeSH Terms: conditions — Dupuytren Contracture | interventions — xiapex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collagenase injection (Active Comparator): Injection of collagenase obtained from Clostridium Histolyticum in contracture string
  Interventions: Drug: Xiapex
- Percutaneous needle fasciotomy (Active Comparator): PNF ad modum Lermusiaux and Debeyre
  Interventions: Procedure: Percutaneous needle fasciotomy

INTERVENTIONS:
Drug: Xiapex — Collagenase Clostridium Histolyticum
  Other Names: XIAPEX® - Pfizer UK
  Arms: Collagenase injection
Procedure: Percutaneous needle fasciotomy — Percutaneous needle fasciotomy ad modum Lermusiaux and Debeyre
  Arms: Percutaneous needle fasciotomy

SUMMARY:
Comparing injectable collagenase and percutaneous needle fasciotomy for Dupuytren's contracture affecting proximal interphalangeal joints. An open label, medico-independent randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* DC affecting PIP joint with Passive Extension Deficit (PED) more than 20 degrees
* Clearly defined strings

Exclusion Criteria:

* Allergies to used medication
* International Normalised Ratio more than 2.0
* Pregnancy and breastfeeding
* Previous treatment for DC in affected finger
* Former inclusion in the study with another string
* Activity in disease at time of study
* PED more than 20 degrees for Metacarpophalangeal or Distal Interphalangeal joint in affected digit

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | 2 years
  Clinical improvement is defined as a contracture reduction 50% or more from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jeppe Lange, M.D., Study Director — Regionshospitalet Silkeborg
Locations (1):
- Center for Planned surgery - Regionalhospital Silkeborg, Silkeborg, Denmark